CLINICAL TRIAL: NCT04333238
Title: Notation Optimization Through Template Engineering
Acronym: NOTE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB00117171
Record Dates: First submitted 2020-03-29; First posted 2020-04-03 (Actual); Last update posted 2023-03-17 (Actual); Status verified 2020-04

CONDITIONS: Clinical Documentation
Keywords: Progress note; Note template; Electronic medical record; Note quality

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard template (Active Comparator): Usual outpatient progress note with standard Subjective Objective Assessment Plan (SOAP) format
  Interventions: Other: Standard progress note template
- New template (Experimental): The assessment and plan section is placed in the beginning, subjective data grouped into the assessment section, and elements not related to the current presentation were deemphasized
  Interventions: Other: New progress note template

INTERVENTIONS:
Other: New progress note template — Residents assigned to document with new progress note template
  Arms: New template
Other: Standard progress note template — Residents assigned to document with standard progress note template
  Arms: Standard template

SUMMARY:
This is a randomized non-blinded controlled trial of a standard note template versus a redesigned note template using a simulated patient encounter and the electronic medical record.

DETAILED DESCRIPTION:
Residents documented the simulated patient encounter using one of two templates. The standard template was based on the usual outpatient progress note. The new template placed the assessment and plan section in the beginning, grouped subjective data into the assessment section, and deemphasized elements not related to the current presentation.

ELIGIBILITY:
Inclusion Criteria:

* Residents who had open visit slots during their outpatient clinic time

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2017-01-20 (Actual); Primary Completion 2017-04-26 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
Note length | Duration of note entry, up to 2 hours
  Note length in line count.
Time to note completion | Duration of note entry, up to 2 hours
  Time to note completion in minutes.
Note evaluation by authors using a likert scale | Immediately after note entry, up to 1 hour
  Likert-scale survey instrument evaluating perceived organization, structure, and efficiency of note.
Note evaluation by reviewers using the Physician Documentation Quality Instrument | Within 1 year
  Physician Documentation Quality Instrument (PDQI-9) - validated note quality scale composed of 9 metrics. 1 is not at all. 5 is extremely.

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy A Epstein, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Outpatient Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
There is no sensitive or protected information. I am able to share any aspect of this trial to whomever would like to know more.
Supporting Information: Study Protocol

REFERENCES:
- [Derived] Epstein JA, Cofrancesco J Jr, Beach MC, Bertram A, Hedian HF, Mixter S, Yeh HC, Berkenblit G. Effect of Outpatient Note Templates on Note Quality: NOTE (Notation Optimization through Template Engineering) Randomized Clinical Trial. J Gen Intern Med. 2021 Mar;36(3):580-584. doi: 10.1007/s11606-020-06188-0. Epub 2020 Sep 8. PMID 32901441